CLINICAL TRIAL: NCT04907279
Title: A Canadian Non-interventional Study of Aripiprazole Once-Monthly (AOM) Administration in Hospitalized Patients With Schizophrenia, Schizoaffective Disorder and Bipolar I Disorder
Brief Title: Aripiprazole Once-Monthly in Hospitalized Patients (INITIATE)
Acronym: INITIATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Otsuka Canada Pharmaceutical Inc. (Industry)
Collaborators: Lundbeck Canada Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-203-00468
Record Dates: First submitted 2021-05-21; First posted 2021-05-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Bipolar I Disorder
Keywords: Aripiprazole; Long-Acting Injectable; Schizophrenia; Schizoaffective Disorder; Bipolar I Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aripiprazole Once-Monthly (AOM) — Dosage and frequency of AOM administration individualized for each study participant in accordance with investigators' clinical judgment.

SUMMARY:
To characterize the real-life clinical use of AOM in a hospitalized patient population with schizophrenia, schizoaffective disorder or BP1 requiring LAI therapy and evaluate its short-term effectiveness associated with its clinical use in the proposed patient population, including time to discharge, efficacy, safety, tolerability, and patients' satisfaction.

DETAILED DESCRIPTION:
This is a non-interventional, Canadian, prospective multi-site study in schizophrenia, schizoaffective disorder and BP1 among in-patients treated with AOM at the discretion of the treating physician and followed for the duration of their hospital stay. With the objective of characterizing the real-life, in-patient clinical uses of AOM, this study will not impose any treatments outside of what is recommended by the attending physician. As such, only patients admitted into hospital and prescribed AOM as a part of their physician's treatment recommendation will be included in this study. Study assessments and administration of questionnaires will be limited to baseline measurements occurring within the first 72 hours of AOM administration and at the end of study participation. All patients will be treated with AOM at the dose that is as per the treating physician's judgment. The decision to treat the patient with AOM must be reached independently and in advance of recruitment in the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is between the age of majority (18 or 19 depending on the province) and 64 years of age inclusively;
2. The patient is currently hospitalized for the treatment of schizophrenia, schizoaffective disorder or BP1;
3. The patient is diagnosed with schizophrenia, schizoaffective disorder, or BP1 as defined by DSM-5 criteria;
4. The treating physician reached the decision to treat the patient with AOM prior to and independently of soliciting the patient to participate in the study;
5. The patient initiated treatment with AOM prior to enrolment and in accordance with routine clinical practice, including the assessment of potential risks associated with the medication (e.g. suicidality);
6. The patient or legal guardian (if applicable and when allowable by law) signed an informed consent indicating the understanding of the study and allowing the use of their anonymous data for the purposes of the study; and
7. The patient and caregiver(s) (if applicable) is/are fluent in English or French, in order to be able to complete the patient-administered questionnaires.

Exclusion Criteria:

1. As per clinical judgement of the treating physician, the patient is diagnosed with treatment-resistant schizophrenia;
2. The patient does not comprehend or refuses to sign the informed consent;
3. The patient is unlikely to comply with study procedures according to the clinical judgment of the investigator;
4. The patient has any contraindications to the use of AOM as specified in the Canadian Product Monograph;
5. The patient is a member of the study personnel or of their immediate families or is a subordinate (or immediate family member of a subordinate) to any of the study personnel;
6. The patient has previously been enrolled in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a primary diagnosis of schizophrenia, schizoaffective disorder or bipolar I disorder requiring hospitalization and for whom, according to the clinical judgment of the treating clinician, Aripiprazole Once-Monthly is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Average dose of Aripiprazole Once Monthly (AOM) | Through study completion, an average of 3 weeks
  The average total dose of AOM administered (number of mg and frequency of administration) during the hospitalization period will be evaluated

SECONDARY OUTCOMES:
Duration of hospital stay | Through study completion, an average of 3 weeks
  Number of days between initiation of AOM and termination of hospital stay
Clinical Global Impression-Improvement (CGI-I) score | Through study completion, an average of 3 weeks
  Mean change in clinical symptom severity from baseline
Global Impression-Severity of Illness (CGI-S) score | Through study completion, an average of 3 weeks
  Mean global severity of clinical symptoms
Personal and Social Performance (PSP) score | Through study completion, an average of 3 weeks
  Mean psycho-social functioning score
Medication Satisfaction Questionnaire (MSQ) score | Through study completion, an average of 3 weeks
  Mean score/level of satisfaction with current treatment administered

CONTACTS AND LOCATIONS:
Overall Officials: Francois Therrien, Pharm.D., Study Director — Otsuka Canada Pharmaceutical Inc.
Locations (1):
- Ottawa Hospital, Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided